CLINICAL TRIAL: NCT06208553
Title: Moving Towards Equity in Hip and Knee Replacement Rehabilitation: A Feasibility Study to Test Implementation of Online Quality Indicator Toolkits
Brief Title: Testing Implementation of Total Joint Replacement Rehabilitation Quality Indicator Toolkits
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of British Columbia (Other)
Collaborators: The Arthritis Society, Canada (Other); Centre for Aging SMART (Unknown); Centre for Advancing Health Outcomes (Unknown)
Responsible Party: Principal Investigator, Marie Westby, Clinical Associate Professor, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: SOG-21-0115)
Record Dates: First submitted 2023-12-18; First posted 2024-01-17 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Arthroplasty, Replacement, Hip; Arthroplasty, Replacement, Knee
Keywords: Rehabilitation; Physical therapy; Quality indicators

STUDY DESIGN:
Intervention Model Description: Single phase (step) of larger stepped-wedge cluster randomized trial design in which 3-month baseline period serves as pre-test after which implementation intervention is introduced (intervention phase) and then post-test data collected (similar to time series design).
Masking Description: Patient and clinician outcome measures are self-reported and therefore not blinded to study phase. Chart auditors will not be blinded to study phase.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: QI toolkit implementation — Patients and clinicians will have access to online toolkits of resources (e.g., video, checklist, rehabilitation tracker, quick guides) reflecting quality indicators for rehabilitation care after total hip and knee replacement surgery.

SUMMARY:
The goal of this feasibility study is to test the procedures for implementing quality indicator toolkits for hip and knee replacement rehabilitation in clinical settings. The main questions it aims to answer are:

* Are the EQUIP (for patients) and QUICK (for clinicians) toolkit resources feasible (accessible, acceptable, usable) in real world clinical settings?
* Are study procedures including recruitment and retention, informed consent, clinical site tracking, audit and feedback, training and data collection feasible?
* What effect does toolkit implementation have on patient experiences, quality of care and patient-reported outcomes? Participants will be asked to provide consent at time of discharge from rehabilitation to have their clinical records audited and to complete an online questionnaire about their physical function, quality of care they received, and overall rehabilitation experience and satisfaction. Rehabilitation providers will also be asked to complete a questionnaire on their adherence to ten post-acute rehabilitation quality indicators after a 3-month baseline period and 6-month implementation phase.

DETAILED DESCRIPTION:
Most people do some form of supervised rehabilitation after hip and knee replacement surgery. Rehabilitation includes assessing pain, mobility, strength, and day-to-day physical function and then prescribing exercises and other interventions to help patients achieve their goals for recovery. Rehabilitation care differs across hospitals, jurisdictions and countries. This can result in some people not receiving the recommended standard of care and not achieving satisfactory outcomes. Study investigators developed 10 quality indicators (QIs) that reflect research-based standards of rehabilitation care after elective hip and knee replacement. The investigators then created a variety of QI resources, in the form of 'toolkits', to share with patients and rehabilitation providers. A feasibility study is being conducted to see if implementing these online toolkits affects the quality and consistency of care patients receive during their rehabilitation at two clinical sites and with up to 135 patients.

As a feasibility study, the investigators are testing the study plan and determining whether enough participants will join a larger study and accept the study procedures.

Clinicians at the two study sites will be asked to:

* Complete a clinician QI questionnaire twice to monitor any change in self-reported adherence to the quality indicators
* Participate in an initial focus group at the start of the 3-month control phase to identify potential barriers and facilitators to using online best practice resources such as QI toolkits and explore the evidence-based practice culture at each site.
* Participate in a 1-hour online training session to introduce QUICK toolkit resources, have questions answered, and receive clinic-level audit and feedback results to better understand any care gaps or areas for improvement.
* Login and access the online QUICK toolkit within the first 3 months of the implementation phase and continue to use throughout the remaining study period. Use of the toolkit is not prescriptive and clinicians can select resources that are most relevant or helpful to them.
* At end of the 9-month study, clinicians will be invited to participate in another focus group meeting to share their views on the toolkits and any challenges to implementing the QIs.
* Throughout the 9-month study, notify the site coordinator when a potentially eligible patient is nearing discharge from their rehabilitation program to facilitate screening and recruitment.

The site-specific clinical champions/site coordinators will provide patients with a postcard with study information and with patient permission, provide contact information to the research assistant. Patients can also opt to contact the study team directly to determine study eligibility and undertake the informed consent process.

Patients at participating sites will be asked to:

* Give consent to have their clinical records (physical therapy notes) audited by trained, independent physical therapy auditors to assess adherence to the quality indicators AND
* Complete an online or paper questionnaire consisting of three separate questionnaires: 1) perception of quality of rehabilitation care; 2) self-reported ability to do every day activities, and 3) rehabilitation experience and satisfaction with care and outcomes. These can be done at home after completion of supervised rehabilitation and will take 15-20 minutes to complete. There is no further follow-up with patients.
* If receiving rehabilitation services after the 3-month control phase, patients will have access to the online EQUIP toolkit (no registration required) and will be encouraged to view resources that are helpful to them for the duration of the study period.

Demographic, clinic and feasibility data will be analyzed descriptively and reported at the clinic level to protect the privacy of participating clinicians. Adherence to the QIs will be examined descriptively and by comparing pooled mean QI adherence pre- and post-implementation using a multiple regression model adjusting for site and baseline patient characteristics: sex, gender, age, surgery (TKR vs THR), co-morbidities, other lower limb involvement, body mass index and education level. Exploratory analysis will include determining level of agreement in QI adherence between data collection tools (e.g., agreement between linked audit tool and patient questionnaire) as well as any signal of quality of care being associated with patient-self reported function and experience. Focus groups will be recorded and transcribed verbatim for thematic analysis and to assist with interpretation of findings.

ELIGIBILITY:
Inclusion Criteria:

Clinician participants

- Physical therapists, rehabilitation assistants, students, and other rehabilitation providers at the study clinical site who provide direct patient care after total joint replacement

Patient participants

* Adults ages 19 and older
* Primary total hip or knee replacement for osteoarthritis
* No significant co-morbidities or peri-operative complications that markedly prolonged acute hospital stay or delayed the start of post-acute rehabilitation
* Sufficient English language skills to provide informed consent and complete questionnaires (with/without help from a family member)
* Completed their course of supervised rehabilitation at study site

Exclusion Criteria:

* Unwilling or unable to provide written informed consent
* Had another lower limb joint replacement in the previous 6 months
* Received some of their post-acute rehabilitation at another clinical facility other than the two study sites
* Received fewer than 3 post-acute rehabilitation visits

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Quality indicator adherence - chart audits | Continuous data collection over 9-month study (through study completion)
  Standardized, purpose-built online audit tool to capture adherence to 10 quality indicators, measured as number of QIs met out of 10, expressed as percentage

SECONDARY OUTCOMES:
Quality indicator adherence - patient questionnaire | Continuous data collection over 9-month study (through study completion)
  Online patient self-report of rehabilitation adherence to 10 quality indicators, measured as number of QIs met out of 10, expressed as percentage
Quality indicator adherence - clinician questionnaire | End of baseline (3 month control period) and end of study (9 months)
  Online clinician self-report of adherence to 10 quality indicators, measured as number of QIs met out of 10, expressed as percentage
Knee injury and Osteoarthritis Outcome Score (KOOS) | Continuous data collection over 9-month study (through study completion)
  Self-reported outcome measures assessing patient's opinion about their pain, other symptoms, daily function and quality of life in past week.
Hip disability and Osteoarthritis Outcome Score (HOOS) | Continuous data collection over 9-month study (through study completion)
  Self-reported outcome measures assessing patient's opinion about their pain, other symptoms, daily function and quality of life in past week.

OTHER OUTCOMES:
Patient rehabilitation experience questionnaire | Continuous data collection over 9-month study (through study completion)
  Study-specific, pilot-tested questionnaire to capture patients' views on overall experience (10 items) and satisfaction with outcomes (8 items) using a 4-point ordinal scale (Not at all, Somewhat, For the most part, Definitely)
Patient feasibility outcomes (patient recruitment rate, consent rate, questionnaire completion rate) | Continuous data collection over 9-month study (through study completion)
  Percentage of patient participants who: are recruited at time of discharge (Denominator: number of TJR patients discharged from clinical site); meet eligibility criteria (Denominator: number screened for participation); provide informed consent (Denominator: number eligible to participate); and complete study questionnaires (Denominator: number sent questionnaires).
Clinician feasibility outcomes (clinician consent rate, training completion rate, toolkit registration rate, focus group participation rate) | Continuous data monitoring over 9-month study (through study completion)
  Percentage of clinician participants who: consent to participate (Denominator: number of eligible clinicians in clinic); complete study training (Denominator: number who consented to participate); register to access QUICK toolkit; (Denominator: number who consented to participate); and participate in baseline and end of study focus groups (Denominator: number who consented to participate).
Toolkit user metrics - page views | Continuous data collection during month 4 to 9 (post-intervention)
  Number of views for each page of the EQUIP and QUICK toolkits.
Toolkit user metrics - average time on page | Continuous data collection during month 4 to 9 (post-intervention)
  Average time spent on each page of the EQUIP and QUICK toolkits.
Toolkit user metrics - page downloads | Continuous data collection during month 4 to 9 (post-intervention)
  Number of times each page was downloaded from the EQUIP and QUICK toolkits.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Aging SMART, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No